CLINICAL TRIAL: NCT04742582
Title: The Potential Protective Effect of a Formula Supplemented With Fermented Matrices on the Risk of Developing Neonatal Sepsis
Brief Title: Potential Protective Effect of a Formula Supplemented With Fermented Matrices on the Risk of Developing Neonatal Sepsis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Heinz Italia SpA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CO-2016-02365100
Record Dates: First submitted 2020-12-31; First posted 2021-02-08 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-06

CONDITIONS: Neonatal Sepsis
MeSH Terms: conditions — Neonatal Sepsis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Preterm Infants - fed fermented formula (Active Comparator): Feeding infants with fermented formula milk. Preterm infants will be fed either with fermented formula milk or with standard formula
  Interventions: Dietary Supplement: Preterm Infants - fed fermented formula
- Preterm Infants - fed standard formula (Placebo Comparator): Feeding infants with standard formula milk. Preterm infants will be fed either with fermented formula milk or with standard formula
  Interventions: Other: Preterm Infants - fed standard formula
- Reference Group: Pre-term Infants - breastfed (Other): The breastfeeding infants were the reference group
  Interventions: Other: Pre-term Infants - breastfed

INTERVENTIONS:
Dietary Supplement: Preterm Infants - fed fermented formula — Feeding infants with fermented formula supplemented with the fermentation products of the probiotic L. paracasei CBA L74 (800 mg / 100 ml of milk) (84 kcal and 2.9 g protein per 100 ml)
  Arms: Preterm Infants - fed fermented formula
Other: Preterm Infants - fed standard formula — Feeding infants with standard formula with the addition of skimmed milk powder in order to provide the same protein and energy amount of the supplemented formula (84 kcal and 2.9 g protein per 100 ml)
  Arms: Preterm Infants - fed standard formula
Other: Pre-term Infants - breastfed — Breastfeeding infants - Reference group
  Arms: Reference Group: Pre-term Infants - breastfed

SUMMARY:
This is a multicenter, randomized, double-blind, placebo controlled trial, with parallel groups and reference group.

The aim of the study was to evaluate the hypothesis that an immunonutritional strategy, based on use of Lactobacillus paracasei CBA L74-fermented formula, prevents or limits the development of late-onset-sepsis in preterm infants.

DETAILED DESCRIPTION:
15-20% of infant born weighing less than 1500 grams develop late-onset-sepsis. The prevention of sepsis is based on hygiene measures, on the prudent use of invasive procedures, on drug management and on early diagnosis. However, no intervention is fully effective in reducing the burden of the disease, prolonged hospitalizations in neonatal intensive care units, high costs or delayed neurodevelopmental impairment. The immunonutrition is defined as the potential to modulate the activity of the immune system throught use of specific nutrients. Many immunonutritional approaches in pediatric age act in part with a modulation of the microbiota. Functional foods derived from fermentation with probiotic strains can be used and their activity is considered specific for each strain and dose dependent.

A new functional food derived from fermentation of cow's milk with Lactobacillus paracasei CBA L74 has recently been de-veloped. The fermentation was started in the presence of 106 bacteria, reaching 5.9 X 109 colony-forming units/g after a 15-h incubation at 37 C°. After heating at 85 C° for 20 s in order to inactivate the live bacteria, the formula was spray-dried. Thus, the final fermented milk powder contained only bacterial bodies and fermentation products and no living microorganisms. Lactobacillus paracasei CBA L74 was registered in the Belgian Collection BCCM/LMG and was included in the EFSA list be-tween the "Qualified Presumption of Safety microorganisms".

Pre-clinical studies showed anti-infective and anti-inflammatory properties of this new fermented food. More recently, a similar effect for the L. paracasei supernatant was noted after 24 and 6 h before the LPS treatment. The supernatant protects against the release of inflammatory mediators IFN-ɣ and IL-12p40 and increases the anti-inflammatory cytokine IL-10.

In a randomized controlled clinical trial, the daily supplementation of this fermented food was shown to protect children from infectious diseases and induces immunoregulatory effects. These clinical results are supported by the significant inverse correlation between the concentrations of alpha-defensins, betadefensins, cathelecidins and the secretory levels of IgA with the number of infectious diseases. In another clinical trial it was shown that a daily supplementation of this new fermented food in healthy full-term infants can stimulate the production of innate and acquired immune peptides. Finally, it was reported that milk fermented by L. paracasei CBA L74 stimultes the immune and non-immune defense mechanisms against sepsis, through a direct interaction with human enterocytes.

Although currently available data suggest a positive impact on morbidity, mortality and costs related to neonatal sepsis, there is little knowledge on the use of this fermented functional food in neonatal age. In particular, there are no studies on the effects of this immunonutritional approach on pre-term infants.

ELIGIBILITY:
Inclusion Criteria:

* Newborns weighing less than 1500 grams
* Gestational age <32 weeks
* Artificial feeding or Human milk not available < 30%

Exclusion Criteria:

* Voluntary interruption;
* Suspension decided by PI or PDF
* Adverse events
* Gastrointestinal disease that prevent oral feeding
* Congenital or maternal infections
* Immunodeficiencies
* Malformations
* Syndromes
* Genetic or metabolic diseases.

Max Age: 72 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 876 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Monitoring of the number of confirmed episodes of late-onset-sepsis during hospitalization period and potential complications of the sepsis | from enrollment (from 0 to 72 hours of life) to discharge (estimated average 40 weeks of corrected age)
  Data collection concerning the appearance during hospitalization of episodes of sepsis from Gram positive, Gram negative bacteria and from fungi; the occurrence of comorbidities: necrotizing enterocolitis (NEC); bronchopulmonary dysplasia (BPD); intraventricular haemorrhage (IVH), retinopathy of prematurity (ROP), the mortality rate.
Monitoring the number of days required to achieve complete enteral feeding, presence and duration of central vascular access | from enrollment (from 0 to 72 hours of life) to discharge (estimated average 40 weeks of corrected age)
  Data collection concerning the number of days required to achieve complete enteral feeding, presence and duration of central vascular access
Monitoring the growth rate | from enrollment (from 0 to 72 hours of life) to discharge (estimated average 40 weeks of corrected age)
  Data collection concerning the growth rate (g/ kg/ day)
Monitoring the length of hospital stay | from enrollment (from 0 to 72 hours of life) to discharge (estimated average 40 weeks of corrected age)
  Data collection concerning the lenght of the hospital stay
Psychomotor development with the Griffiths III | at 180 days of life
  Evaluation of the psychomotor development through development quotient using the Griffiths III. General quotient: A scale: learning basis; B scale: language and communication; C scale: eye-manual coordination; D scale: personal-social-emotional; E scale: gross-motor; average 100, DS 15.

SECONDARY OUTCOMES:
Fecal dosage of cathelicidines, alfa and beta defensins, sIgA | at the enrollment (from 0 to 72 hours of life), at 30 days of life, and discharge or 40 weeks of correct age
  Dosage of biomarkers levels of innate and acquired immunity (cathelicidines, alfa and beta defensins, sIgA ) on fecal samples, using ELISA kits
Microbiota | at the enrollment (from 0 to 72 hours of life), at 30 days of life, and discharge or 40 weeks of correct age
  The V region of the 16S rRNA will be amplified using specific primers and the obtained amplicons will be used for sequencing library preparation, multiplexing and paired-end sequencing on the Illumina MiSeq platform. The alpha and beta diversity at the level of the phylum, genus and species among groups and their separation in a principal coordinate analysis will be evaluated.
Cytokines production assessment on infants blood sample | at the enrollment (from 0 to 72 hours of life), at 30 days of life, and discharge or 40 weeks of correct age
  Cytokines (IL-6, IL-12p40, TNF-a) production assessment on infants blood sample, using CBA (cytokine bead array)
Cytokines production assessment on dendritic cells culture medium | at the enrollment (from 0 to 72 hours of life), at 30 days of life, and discharge or 40 weeks of correct age
  Cytokines (IL-6, IL-12p40, TNF-a) production assessment on murine dendritic cells culture medium
Cell surface activation markers (MHC and costimulatory molecules) | at the enrollment (from 0 to 72 hours of life), at 30 days of life, and discharge or 40 weeks of correct age
  Determination of cell surface activation markers (MHC and costimulatory molecules) on dendritic cell after infant serum treatment and strong inflammatory stimulus (LPS or Salmonella typhimurium)

CONTACTS AND LOCATIONS:
Locations (1):
- Unità di Neonatologia e Terapia Intensiva Neonatale, Clinica Mangiagalli, Milan, Italy